CLINICAL TRIAL: NCT02665832
Title: A Randomized, Open-label, Single-Dose, 2-Way Cross-over Study To Compare the Safety and Pharmacokinetic Characteristics of Combination of Amlodipine, Olmesartan and Rosuvastatin and DWJ1351 in Healthy Male Volunteers
Brief Title: Study of DWJ1351 in Healthy Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DW_DWJ1351002
Record Dates: First submitted 2016-01-20; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — olmesartan; Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AB (Experimental): Sevikar (Olmesartan/Amlodipine) and Crestor (Rosuvastatin) followed by DWJ1351
  Interventions: Drug: DWJ1351; Drug: Co-administration of Sevikar (Olmesartan/Amlodipine) and Crestor (Rosuvastatin)
- BA (Experimental): DWJ1351 followed by Sevikar (Olmesartan/Amlodipine) and Crestor (Rosuvastatin)
  Interventions: Drug: DWJ1351; Drug: Co-administration of Sevikar (Olmesartan/Amlodipine) and Crestor (Rosuvastatin)

INTERVENTIONS:
Drug: DWJ1351
Drug: Co-administration of Sevikar (Olmesartan/Amlodipine) and Crestor (Rosuvastatin)

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetic characteristics of combination of amlodipine, olmesartan and rosuvastatin and DWJ1351 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male subjects aged 19 to 50 years
* Subjects whose body weight ≥ 55 kg and Body Mass Index(BMI) ≥ 18.0 kg/m2 and ≤ 27.0 kg/m2
* Subject who was judged to be healthy and suitable for the participation by the investigator based on screening test results
* Subject who provided written informed consent to participate in this study

Exclusion Criteria:

* Subject who had a severe allergy or allergic reactions to the amlodipine, olmesartan, rosuvastatin or related drugs
* Subject with sign or symptoms or previously diagnosed disease of liver, kidney, neurology, respiratory, endocrinology, hematology, cardiovascular, digestive system, reproductive system, neurology, psychology, ophthalmic and skin disease
* Subjects who had a serious clinical illness that can impact fate of drugs absorption
* Subject who shows vital signs with the number of systolic blood pressure of ≥150 mmHg or ≤100 mmHg, and the number of diastolic blood pressure of ≥100mmHg or ≤66mmHg
* Subject who have experienced drug abuse
* Subject who donates his blood (whole blood donation within last 2 months or plasma donation within last 1 month)
* Subject who has taken other clinical or licensed medication from another clinical trial within an 3-month period prior to the first administration of the study medication

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
AUC | 0 - 144 hr
Cmax | 0 - 144 hr